CLINICAL TRIAL: NCT03414216
Title: Surgical Offloading Procedures for Diabetic Foot Ulcers Compared to Best Non-surgical Treatment
Brief Title: Surgical Offloading Procedures for Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf Harofeh MC (Other Government)
Responsible Party: Sponsor-Investigator, Assaf Harofeh MC, Senior Orthopaedic Surgeon, Assaf-Harofeh Medical Center
Organization: Assaf-Harofeh Medical Center (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0094-17-ASF
Record Dates: First submitted 2017-12-22; First posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot | interventions — Casts, Surgical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 - early off-loading surgery (Experimental): Within 1 week of randomization, offloading surgery:
  Tip of toe ulcers will be treated by percutaneous tenotomy. Ulcers under metatarsal heads will be offloaded with minimally invasive floating metatarsal osteotomy.
  Ulcers plantar to the interphalangeal joint of the hallux will be treated by a modified Keller resection arthroplasty.
  Interventions: Procedure: Group 1 early offloading surgery
- Group 2 - off-loading in fiberglass cast (Active Comparator): Tip of toe ulcers and ulcers plantar to the interphalangeal joint of the big toe will be casted in a fiberglass cast with a heel, ending under the metatarsal heads, leaving the toes in the air.
  Ulcers under metatarsal heads will be casted in a full foot fiberglass cast with a heel with a window below the ulcer designed to relieve pressure under the metatarsal heads.
  Interventions: Procedure: Group 2 - off-loading in fiberglass cast

INTERVENTIONS:
Procedure: Group 1 early offloading surgery — As above.
  Arms: Group1 - early off-loading surgery
Procedure: Group 2 - off-loading in fiberglass cast — As above.
  Arms: Group 2 - off-loading in fiberglass cast

SUMMARY:
100 consenting subjects with Texas grade 1a diabetic foot ulcers will be randomized to surgical offloading or non-operative offloading.

DETAILED DESCRIPTION:
Background: Diabetic foot ulcers are frequently related to elevated pressure under a bony prominence. Conservative treatment includes offloading with orthopaedic shoes and custom made orthotics or plaster casts. While casting in plaster is usually effective in achieving primary closure of foot ulcers, recurrence rates are high. Minimally invasive surgical offloading that includes correction of foot deformities has good short and long term results. The surgery alleviates the pressure under the bony prominence, thus enabling prompt ulcer healing, negating the patient's dependence on expensive shoes and orthotics, with a lower chance of recurrence. The purpose of this protocol is to compare offloading surgery (percutaneous flexor tenotomy, mini-invasive floating metatarsal osteotomy or Keller arthroplasty) to non-surgical treatment for patients with diabetic foot ulcers in a crossover designed RCT.

Methods: 100 patients with diabetic neuropathy related foot ulcers (tip of toe ulcers, ulcers under metatarsal heads and ulcers under the hallux interphalangeal joint) will be randomized (2:3) to a surgical offloading procedure or best available non-surgical treatment. Group 1 (surgery) will have surgery within 1 week. Group 2 (controls) will be prescribed an offloading cast applied for up to 12 weeks (based on clinical considerations). Following successful offloading treatment (ulcer closure with complete epithelization) patients will be prescribed orthopaedic shoes and custom made orthotics. If offloading by cast for at least 6 weeks fails, or the ulcer recurs, patients will be offered surgical offloading. Follow-up will take place till 2 years following randomization. Outcome criteria will be time to healing of the primary ulcer (complete epithelization), time to healing of surgical wound, recurrence of ulcer, time to recurrence and complications.

Discussion: The high recurrence rate of foot ulcers and their dire consequences justify attempts to find better solutions that the non-surgical options available at present. To promote surgery, randomized controlled trial (RCT) level evidence of efficacy is necessary.

ELIGIBILITY:
Inclusion Criteria:

* Single Texas A1 or A2 ulcer.
* ulcer attributable to an anatomic deformity.

Exclusion Criteria:

* Unable to understand language of informed consent.
* Ischemia.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Failure to cure | 12 weeks
  Lack of full epithelization
Any recurrence of any ulcer at same location | 2 years
  If either of the outcomes is positive, the case will be counted as a failure.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Finestone AS, Tamir E, Ron G, Wiser I, Agar G. Surgical offloading procedures for diabetic foot ulcers compared to best non-surgical treatment: a study protocol for a randomized controlled trial. J Foot Ankle Res. 2018 Feb 20;11:6. doi: 10.1186/s13047-018-0248-3. eCollection 2018. PMID 29467829